CLINICAL TRIAL: NCT02687399
Title: A Phase II/III, Randomized, Controlled, Single Blind Study to Evaluate the Haemostatic Efficacy and Safety of Topically Applied TT-173 in Patients Undergoing Knee Arthroplasty
Brief Title: Determine the Efficacy of TT-173. Reducing the the Total Blood Loss Associated With Total Knee Arthroplasty (HESTAT)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thrombotargets Europe S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THO-IM_02-CT; 2015-003408-21 (EudraCT Number)
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Degenerative Osteoarthritis
Keywords: knee arthroplasty
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TT-173 (Experimental): It will be sprayed using this syringe and a nozzle tip couplet to it one time over the surgical lesion surfaces on the exposed tissues of the knee
  Interventions: Biological: TT-173
- placebo (Placebo Comparator): It will be sprayed over the surgical lesion surfaces on the exposed tissues of the knee
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — After prosthesis cementation and just before knee suture and tourniquet liberation, the patients randomized in the placebo group will receive placebo for inyection sprayed on the exposed tissues of the knee.
  Arms: placebo
Biological: TT-173 — After prosthesis cementation and just before knee suture and tourniquet liberation, the patients randomized in the treatment group will receive TT-173 for inyection sprayed on the exposed tissues of the knee.
  Arms: TT-173

SUMMARY:
The purpose of this study is to determine the haemostatic efficacy of TT-173, reducing the total blood loss associated with the total knee arthroplasty.

DETAILED DESCRIPTION:
As the TT-173 has been cleared for use as a topical hemostatic agent, the proposed study will further investigate the safety and efficacy of TT-173 in the knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who signed the informed consent.
2. Patients affected of degenerative osteoarthritis of the knee that have to undergo a primary total knee replacement.
3. Patients of both sexes older than 18 years.
4. Female patients in childbearing age* that are not permanently sterile, should present a negative pregnancy test and should agree to use a medically accepted anti contraceptive method during its participation in the study. This includes oral, intravaginal, transdermal, injectable or implantable hormonal contraceptives, sexual abstinence, bilateral tubal occlusion, intrauterine hormone-releasing system or dispositive and vasectomy of the partner.

   * Includes the period between menarche and until becoming post-menopausal. A woman is considered post-menopausal when she has gone without a period for 12 consecutive months.
5. Patients must have a haemoglobin concentration ≥ to 12.5 g/dL at the selection visit.

Exclusion Criteria:

1. Patients affected of any kind of congenital or acquired coagulopathies or with personal history of abnormal haemorrhagic episodes.
2. Patients subjected to knee replacement due to rheumatoid or seronegative arthritis, infection or other autoimmune inflammatory causes of join degeneration.
3. Patients subjected to revision procedures of the knee, hemiarthroplasty or that will receive non-cemented knee prosthesis.
4. Subjects affected of a serious medical condition that would compromise their clinical outcome such as hepatic, respiratory, cardiac or renal insufficiency, acute infectious disease and active cancer.
5. Subjects with known history of haematological alterations which are causative of thrombophilia.
6. Subjects with personal history of deep vein thrombosis, pulmonary thromboembolism, retinal vascular occlusion or multiple abortions.
7. Subjects with known hypersensitivity or allergy to any component of the drug.
8. Subjects that are currently under treatment with anticoagulant, antiplatelet or antifibrinolytic drugs. These subjects may be eligible if the treatment is stopped preoperatively according with the conditions indicated in section 9.2.
9. Subjects who have received treatment (erythropoietin, iron, folate) to improve preoperative anaemia.
10. Subjects who are not free to give informed consent or who are mentally incapacitated to the discretion of investigators.
11. Subjects who participate or have participated in the past three months in another clinical trial with drug treatment.
12. Subjects that are the investigators, collaborators, nurses, centre employees or any other person directly related to the development of the protocol.
13. Subjects who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
total blood loss | 2 day

SECONDARY OUTCOMES:
Maximum decrease in venous haemoglobin concentration | 2 day
Blood collected in the drainage | 1 day
Transfusion rate | 35 days
Number of units of blood concentrates transfused | 35 days
Range of knee motion (Knee flexion and extension) | 35 days
Systemic absorption (detectable increase of TF blood concentration at any time of the pharmacokinetics sampling) | 15 days
Immunogenicity (detectable increase of reactive antibodies against the product ) | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Rojas, Study Director — Thrombotargets Europe
Locations (1):
- Thrombotargets Europe SL, Castelldefels, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lopez-Lopez J, Jane-Salas E, Santamaria A, Gonzalez-Navarro B, Arranz-Obispo C, Lopez R, Miquel I, Arias B, Sanchez P, Rincon E, Rodriguez JR, Rojas S, Murat J. TETIS study: evaluation of new topical hemostatic agent TT-173 in tooth extraction. Clin Oral Investig. 2016 Jun;20(5):1055-63. doi: 10.1007/s00784-015-1586-1. Epub 2015 Sep 15. PMID 26374745
- [Derived] Gonzalez-Osuna A, Videla S, Canovas E, Urrutia G, Rojas S, Lopez R, Murat J, Aguilera X. HESTAT: Study protocol for a phase II/III, randomized, placebo-controlled, single blind study to evaluate the new hemostatic agent TT-173 in total knee arthroplasty. Contemp Clin Trials. 2017 Oct;61:16-22. doi: 10.1016/j.cct.2017.07.004. Epub 2017 Jul 4. PMID 28687347
- See also: For more information about this study; Clinical Oral Investigations journal — http://link.springer.com/article/10.1007%2Fs00784-015-1586-1